CLINICAL TRIAL: NCT04951765
Title: A Phase I Study to Examine the Effects of Low and High-fat Meals on Orally Administered XZP-3287 in Healthy Adult Subjects
Brief Title: Effect of Food on the Pharmacokinetics of XZP-3287 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: XZP-3287-1002
Record Dates: First submitted 2021-06-16; First posted 2021-07-07 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-06

CONDITIONS: Healthy
Keywords: XZP-3287; Food Effect; Pharmacokinetics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm A (Experimental): Cycle1 Day 1：fasting；Cycle2 Day 1：high-fat meal；Cycle3 Day 1：low-fat meal
  Interventions: Drug: XZP-3287
- Arm B (Experimental): Cycle1 Day 1：high-fat meal；Cycle2 Day 1：low-fat meal；Cycle3 Day 1：fasting
  Interventions: Drug: XZP-3287
- Arm C (Experimental): Cycle1 Day 1：low-fat meal；Cycle2 Day 1：fasting；Cycle3 Day 1：high-fat meal
  Interventions: Drug: XZP-3287
- Arm D (Experimental): Cycle1 Day 1：fasting；Cycle2 Day 1：low-fat meal；Cycle3 Day 1：high-fat meal
  Interventions: Drug: XZP-3287
- Arm E (Experimental): Cycle1 Day 1：high-fat meal；Cycle2 Day 1：fasting；Cycle3 Day 1：low-fat meal
  Interventions: Drug: XZP-3287
- Arm F (Experimental): Cycle1 Day 1：low-fat meal；Cycle2 Day 1：high-fat meal；Cycle3 Day 1：fasting
  Interventions: Drug: XZP-3287

INTERVENTIONS:
Drug: XZP-3287 — Cycle1 Day 1: one dose of XZP-3287 before starting a low-fat breakfast Cycle2 Day 1: one dose of XZP-3287 after finishing a high-fat breakfast Cycle3 Day 1: one dose of XZP-3287 after finishing a low-fat breakfast
  Arms: Arm A
Drug: XZP-3287 — Cycle1 Day 1: one dose of XZP-3287 after finishing a high-fat breakfast Cycle2 Day 1: one dose of XZP-3287 after finishing a low-fat breakfast Cycle3 Day 1: one dose of XZP-3287 before starting a low-fat breakfast
  Arms: Arm B
Drug: XZP-3287 — Cycle1 Day 1: one dose of XZP-3287 after finishing a low-fat breakfast Cycle2 Day 1: one dose of XZP-3287 before starting a low-fat breakfast Cycle3 Day 1: one dose of XZP-3287 after finishing a high-fat breakfast
  Arms: Arm C
Drug: XZP-3287 — Cycle1 Day 1: one dose of XZP-3287 before starting a low-fat breakfast Cycle2 Day 1: one dose of XZP-3287 after finishing a low-fat breakfast Cycle3 Day 1: one dose of XZP-3287 after finishing a high-fat breakfast
  Arms: Arm D
Drug: XZP-3287 — Cycle1 Day 1: one dose of XZP-3287 after finishing a high-fat breakfast Cycle2 Day 1: one dose of XZP-3287 before starting a low-fat breakfast Cycle3 Day 1: one dose of XZP-3287 after finishing a low-fat breakfast
  Arms: Arm E
Drug: XZP-3287 — Cycle1 Day 1: one dose of XZP-3287 after finishing a low-fat breakfast Cycle2 Day 1: one dose of XZP-3287 after finishing a high-fat breakfast Cycle3 Day 1: one dose of XZP-3287 before starting a low-fat breakfast
  Arms: Arm F

SUMMARY:
This study will be a randomized 3-treatment, cross-over study to evaluate the bioavailability of XZP-3287 administered after a high or low-fat meal.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

1. Healthy male or female subjects aged 18 to 65 years (including 18 and 65);
2. Male body weight ≥50kg, female body weight ≥45kg, body mass index between 18 to 28 kg/m2 (inclusive).
3. No medical history of important primary organ diseases such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and musculoskeletal system.
4. Subjects shall ake effective contraceptive measures voluntarily within 3 months from the date of signing the informed consent form (for women, 2 weeks before trial screening) to the date of the last medication.
5. Willing and able to comply with all scheduled visits, study procedures, and provides written informed consent

Exclusion Criteria:

1. Allergic constitution and those with known allergy to XZP-3287 or similar drugs and excipients
2. Abnormal clinical tests and clinical significance judged by the investigator
3. Frequent use of sedatives, sleeping pills or other addictive drugs within 6 months before enrollment
4. History of drug use, or drug abuse screening positive
5. Those who had smoked more than 5 cigarettes per day on average in the 3 months before the screening period or habitually used nicotine-containing products and were unable to quit during the test period
6. Heavy drinking or regular drinking in the six months preceding the screening period
7. Use of any prescription drug or Chinese herbal medicine within 4 weeks prior to enrollment, or use of any over-the-counter drug, any vitamin product, health care drug within 14 days prior to enrollment;
8. Treatment with an investigational drug within 3 months
9. Participated in blood donation with blood donation volume ≥400 mL or received blood transfusion within 3 months before screening.
10. Had a severe infection, trauma or major surgery within 4 weeks of screening
11. Gastrointestinal disorders causing clinically significant symptoms such as nausea, vomiting, and diarrhea, or malabsorption syndromes
12. Pregnant or lactating women, or subjects cannot take strict contraceptive measures as required.
13. Hepatitis B surface antigen or E antigen, hepatitis C antibody, HIV antibody and syphilis antibody, any of which are positive.
14. Allergic to any food ingredients or has special requirements on diet, cannot follow the unified diet
15. habitual consumption of food or beverage containing methylxanthine, such as tea, coffee, cola, chocolate and so on during the study period
16. habitual consumption of grapefruit juice during the study period
17. have difficulty in blood collection or cannot tolerate vein puncture for blood collection
18. As determined by the investigator, the subject has other factors that are not suitable for the study -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Primary PK Endpoints | day 1~day 21
  Cmax
Primary PK Endpoints | day 1~day 21
  AUC0-∞
Primary PK Endpoints | day 1~day 21
  AUC0-t

SECONDARY OUTCOMES:
Secondary PK measures | day 1~day 21
  Tmax
Secondary PK measures | day 1~day 21
  T1/2
Secondary PK measures | day 1~day 21
  CL/F
Secondary PK measures | day 1~day 21
  Vz/F
Safety and tolerability | Up to 14 days after last dose
  Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China